CLINICAL TRIAL: NCT04831658
Title: A Prospective Clinical Study of a New Generation of BTK Inhibitors Combined With PD-1 and Formustine in the First-line Treatment of Primary Central Nervous System Lymphoma
Brief Title: A Prospective Clinical Study of BTK Inhibitor, PD-1 and Formustine in the First-line Treatment of Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20210303
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: BTK inhibitor; PD-1; fotemustine; CRR; ORR; DCR; PFS; OS; ADR; Adverse events; ECOG score; laboratory examination; vital signs; physical examination; Time to disease progression (TTP); median survival (MST); quality of life (QOL); adverse reactions (ADR)
MeSH Terms: conditions — Myeloproliferative Syndrome, Transient

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib combined with PD-1 and fotemustine (Experimental): To observe the efficacy and safety of a new generation of BTK inhibitor abutinib combined with PD-1 and formustine in the treatment of newly-treated patients with primary central nervous system lymphoma (PCNSL)
  Interventions: Drug: the dose-escalation phase

INTERVENTIONS:
Drug: the dose-escalation phase — The study adopts the "3+3" design,The dose planned to be explored is the daily oral dose of the BTK inhibitor abutinib, which is 100 mg, 150 mg and 200 mg, respectively.Orelabrutinib continues to be taken orally until the tumor is relieved for 3 months; PD-1 monoclonal antibody is used by intravenous drip, 21 days as a treatment cycle, and a total of 1 year of observation; formustine is used by intravenous drip for 21 days It is a treatment cycle, a total of 6 cycles of observation; after 2 cycles, the efficacy is evaluated, and adverse reactions are recorded. At the same time, MTX 12mg+Ara-C 50mg+Dex 5mg was injected into the CSF cytology-positive sheath, and intrathecal injection once per treatment cycle, a total of 6 times.
  Other Names: The extended treatment phase

SUMMARY:
To observe the efficacy and safety of a new generation of BTK inhibitor Orelabrutinib combined with PD-1 and fotemustine in the treatment of patients with primary central nervous system lymphoma (PCNSL).

DETAILED DESCRIPTION:
This study includes a dose escalation phase and an extended treatment phase . The dose-escalation phase： Primary study endpoint: Safety endpoint: including dose-limiting toxicity (DLT), adverse events, ECOG performance score, laboratory tests, vital signs, physical examination .

Secondary research endpoints: effectiveness endpoints: including complete response rate (CRR), objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS).

The study adopts the "3+3" design, that is, 3-6 subjects in each group complete the administration, and the dose group determined as the maximum tolerated dose (MTD) is included in the group of 6 subjects, totaling 9-18 example. The dose planned to be explored is the daily oral dose of the BTK inhibitor abutinib, which is 100 mg, 150 mg and 200 mg, respectively. The doses of other drugs in the plan will not be escalated.

After the last subject in each dose group completes the 28-day restricted toxicity (DLT) assessment window after the administration, the investigator can start the entry into the next dose group after evaluating and agreeing to enter the next dose group based on clinical safety data.DLT was defined as any grade 3 or higher nonhematologic toxicity, any grade 4 hematologic toxicity, grade 3 febrile neutropenia, and grade 3 thrombocytopenia with significant bleeding.

When 1 case of DLT occurs among 3 subjects in a certain dose group, 3 subjects need to be added to the same dose group (6 subjects in this dose group complete the DLT assessment): If the additional 3 subjects are tested If there is no DLT, continue the dose escalation; if 1 of the 3 increased subjects has DLT, stop the dose escalation; if the increased 3 subjects have >1 of the subjects DLT, the dose escalation is stopped, and the dose needs to be lowered to continue to enroll 3 subjects for DLT evaluation. If DLT occurs in 2 of the 3 or 6 subjects in the dose group, then the previous low dose is defined as the maximum tolerated dose (MTD).

The extended treatment phase :

Primary study endpoints: objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), overall survival (OS) .

Secondary endpoints: time to disease progression (TTP), median survival (MST), adverse reactions (ADR), quality of life (QOL) .

The study adopts an open, one-arm, prospective clinical collaborative study . The initial treatment is BTK inhibitor (Obutinib), PD-1 monoclonal antibody combined with formustine ：Orelabrutinib continues to be taken orally until the tumor is relieved for 3 months; PD-1 monoclonal antibody is used by intravenous drip, 21 days as a treatment cycle, and a total of 1 year of observation; formustine is used by intravenous drip for 21 days It is a treatment cycle, a total of 6 cycles of observation; after 2 cycles, the efficacy is evaluated, and adverse reactions are recorded. At the same time, MTX 12mg+Ara-C 50mg+Dex 5mg was injected into the CSF cytology-positive sheath, and intrathecal injection once per treatment cycle, a total of 6 times.

Second stage treatment ：The efficacy was evaluated after 6 cycles of treatment in the initial stage. The CR patients continued to take orally abutinib (150mg, qd) for three months, and the PD-1 monoclonal antibody was used for maintenance treatment for up to 1 year; the PR patients received whole brain radiotherapy (WBRT), and at the same time Continue oral obritinib (150mg, qd) for three months and PD-1 monoclonal antibody maintenance treatment for up to one year; SD and PD patients choose methotrexate + pemetrexed combined chemotherapy for 4 cycles followed by whole brain radiotherapy (WBRT). WBRT: Regardless of age, supplementary WBRT 30-36Gy + partial reduction field irradiation up to 45Gy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years; KPS score ≥ 60 points or ECOG score ≤ 2 points; expected survival time of more than 3 months; PCNSL confirmed pathologically by tissue biopsy (limited to the brain, not accompanied by lymphoma in other parts of the body) , And histopathological type is diffuse large B-cell lymphoma; no chemotherapy contraindications (blood picture and physiological examination result time <7 days); at least one measurable lesion according to RECIST standards; no other serious diseases that conflict with this plan ; Follow-up is possible; other anti-tumor drugs are not used during this treatment period, and bisphosphonate anti-bone metastasis therapy and other symptomatic treatments can be applied; understand the situation of this study and sign the informed consent.

Exclusion Criteria:

* Those who are currently receiving other chemical, radiotherapy and targeted therapies (received chemotherapy within 3 weeks, received radiotherapy within 2 weeks, or have not recovered from the acute toxicity of any previous treatment); pregnant or lactating women; yes Any uncontrollable medical disease (including active infection, uncontrolled diabetes, severe heart, liver, kidney dysfunction, and interstitial pneumonia, etc.); those who are contraindicated with chemotherapy such as cachexia; have had other malignant tumors in the past Those who have uncontrolled infections; those who have a history of uncontrollable mental illness; those who are considered unsuitable to participate in this trial by the investigator.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
DLT | up to 24 months
  Dose-limiting toxicity
AE | up to 24 months
  adverse events
ECOG performance score | up to 24 months
  ECOG performance score
laboratory tests | up to 24 months
  laboratory tests
vital signs | up to 24 months
  vital signs
physical examination | up to 24 months
  physical examination
ORR | up to 24 months
  Objective Responder Rate
DCR | up to 24 months
  Disease Control Rate
PFS | up to 24 months
  Progression Free Survival
OS | up to 24 months
  Overall Survival

SECONDARY OUTCOMES:
ORR | up to 24 months
  Objective Responder Rate
DCR | up to 24 months
  Disease Control Rate
PFS | up to 24 months
  Progression Free Survival
OS | up to 24 months
  Overall Survival
ADR | up to 24 months
  Adverse Reaction Rate
CRR | up to 24 months
  complete response rate
TTP | up to 24 months
  Time to disease progression
MST | up to 24 months
  median survival
ADR | up to 24 months
  adverse reactions
QOL | up to 24 months
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Zhao W, Li L, Fu X, Chang Y, Sun Z, Zhu L, Li X, Wang X, Yan J, Jia S, Ma S, Fan M, Qian S, Zhang Y, Yang Q, Qiao H, Chen Q, Zhang M, Zhang X. A first-line regimen combining Bruton's tyrosine kinase and programmed cell death protein-1 inhibitors with chemotherapy excluding methotrexate achieves high response rates in primary central nervous system lymphoma. Cancer. 2026 Jan 1;132(1):e70247. doi: 10.1002/cncr.70247. PMID 41485126